CLINICAL TRIAL: NCT01056744
Title: Endothelial Stent Coverage and Neointimal Proliferation at 6 Months After Implantation of a Coronary Everolimus-Eluting Stent Compared With a Bare Metal Stent Postdilated With a Paclitaxel-Eluting Balloon: A Randomised Study Using Optical Coherence Tomography
Brief Title: Optical Coherence Tomography to Evaluate Paclitaxel-Eluting Balloons and Everolimus-Eluting Coronary Stents
Acronym: OCTOPUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: B. Braun Melsungen AG (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Tudor C. Poerner, PD Dr. med., University of Jena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKJ-TCP-1
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Stents; Neointimal Proliferation
Keywords: coronary stent; optical coherence tomography; drug-eluting; neointimal proliferation
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DES (Active Comparator): Implantation of a XIENCE® V everolimus eluting coronary stent (drug-eluting stent, DES)
  Interventions: Device: Percutaneous coronary intervention with stent implantation
- BMS/DEB (Active Comparator): Implantation of a Coroflex Blue® coronary stent (bare metal stent, BMS) postdilated with a Sequent Please® paclitaxel-eluting balloon (drug-eluting balloon, DEB)
  Interventions: Device: Percutaneous coronary intervention with stent implantation

INTERVENTIONS:
Device: Percutaneous coronary intervention with stent implantation — Percutaneous coronary intervention with implantation of either:
  - a XIENCE® V everolimus eluting coronary stent in one of the following sizes: 3.0 x 18 mm, 3.0 x 28 mm, 2.5 x 18 mm, 2.5 x 28 mm (DES group),
  or:
  - a Coroflex Blue® coronary stent postdilated with a Sequent Please® paclitaxel-eluting balloon in one of the following size combinations (stent / balloon): 3.0 x 16 mm / 3.0 x 20 mm, 3.0 x 25 mm / 3.0 x 30 mm, 2.5 x 16 mm / 2.5 x 20 mm, 2.5 x 25 mm / 2.5 x 30 mm (BMS/DEB group)
  Other Names: XIENCE® V, Coroflex Blue®, Sequent Please®

SUMMARY:
Background:

Safety concerns regarding use of drug eluting stent systems (DES) are related mostly to late stent thrombosis, which is facilitated by incomplete stent endothelial coverage. Specific information about time course and amount of endothelial strut coverage of different DES is required, in order to further refine the concept of antiplatelet therapy after DES implantation. Optical coherence tomography (OCT) is emerging as a new gold standard for endovascular imaging of stents, atherosclerosis progression, vulnerable plaque and neointimal proliferation. Very limited OCT data about endothelial coverage of DES are currently available. Aim of this study is a comparative evaluation of XIENCE V® everolimus eluting stent (Abbot Vascular) and of the bare metal stent (BMS) Coroflex® Blue postdilated with the drug-eluting balloon (DEB) SeQuent® Please (paclitaxel-eluting balloon, B. Braun Melsungen AG) in terms of endothelial coverage and neointimal proliferation using OCT.

Study Design:

A number of 80 patients scheduled for elective percutaneous coronary intervention (PCI) with a native coronary stenosis suitable for DES implantation and OCT imaging are openly randomized 1:1 to either XIENCE V® or Coroflex® Blue/Sequent® Please. The study is prospectively conducted at a university high-volume PCI center with OCT expertise (Jena, Germany). Angiographic follow-up and OCT imaging with motorized pull-back at 1 mm/s are planned in all patients 6 months after implantation of the study stents. OCT endpoints are: (1) endothelial coverage, expressed as % of struts without coverage and % of stent length containing non-covered struts, and respectively (2) neointimal proliferation, given as % neointimal volumetric proliferation within the whole stent and also as focal peak % neointimal area proliferation. The study is not powered for clinical endpoints, which are: subacute or late stent thrombosis and need for revascularization of the stent segment. Given the high number of measurements (15 cross-section images / 1 mm stent length), OCT endpoints are likely to reach significance at the level P < 0.05 even at a follow-up drop-out rate up to 20%.

ELIGIBILITY:
Inclusion Criteria:

* Established indication to PCI according to the guidelines of American Heart Association and American College of Cardiology
* Age > 18 years, written consent
* Native coronary lesion suitable for stent placement and OCT imaging

Exclusion Criteria:

1. General exclusion criteria:

   * Pregnancy and breast feeding mother
   * Co-morbidity with an estimated life expectancy of < 50 % at 1 year
   * Scheduled major surgery in the next 6 months
   * Not able to give informed written consent or non-compliance
   * Participation in other PCI trial
2. Procedural exclusion criteria:

   * Acute coronary syndromes and cardiogenic shock
   * Previous subacute or late coronary stent thrombosis
   * Known non-responsiveness / allergy to aspirin or thienopyridines
   * Known allergy against everolimus or against taxol derivates
3. Angiographic exclusion criteria:

   * Culprit lesion within the proximal 10 mm of the right or left coronary artery
   * Saphenous vein grafts
   * Estimated stent length > 30 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Endothelial coverage of the stent struts assessed by optical coherence tomography | 6 months

SECONDARY OUTCOMES:
Neointimal proliferation within the stent assessed by optical coherence tomography | 6 months
Subacute or late thrombosis of the study stent | 6 months
Need for revascularization of the vessel segment containing the study stent | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tudor C Poerner, MD, PhD, Study Director — Jena University Hospital; Hans R Figulla, Professor, Study Chair — Jena University Hospital
Locations (1):
- University Hospital of Jena, 1st Medical Department, Division of Cardiology, Jena, Germany

REFERENCES:
- [Derived] Poerner TC, Otto S, Gassdorf J, Nitsche K, Janiak F, Scheller B, Goebel B, Jung C, Figulla HR. Stent coverage and neointimal proliferation in bare metal stents postdilated with a Paclitaxel-eluting balloon versus everolimus-eluting stents: prospective randomized study using optical coherence tomography at 6-month follow-up. Circ Cardiovasc Interv. 2014 Dec;7(6):760-7. doi: 10.1161/CIRCINTERVENTIONS.113.001146. Epub 2014 Nov 4. PMID 25371536
- [Derived] Poerner TC, Otto S, Gassdorf J, Janiak F, Danzer C, Ferrari M, Figulla HR. A prospective randomised study using optical coherence tomography to assess endothelial coverage and neointimal proliferation at 6-months after implantation of a coronary everolimus-eluting stent compared with a bare metal stent postdilated with a paclitaxel-eluting balloon (OCTOPUS Trial): rationale, design and methods. EuroIntervention. 2011 May;7 Suppl K:K93-9. doi: 10.4244/EIJV7SKA16. PMID 22027737